CLINICAL TRIAL: NCT02988804
Title: Effects on the Awakening With Laryngeal Mask vs Endotracheal Tube in Endoscopic Endonasal Transsphenoidal Base Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Ricard Valero, MD, PhD, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCB.2016.0781
Record Dates: First submitted 2016-12-01; First posted 2016-12-09 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Skull Base Neoplasms
Keywords: endoscopic endonasal transsphenoidal surgery; laryngeal mask
MeSH Terms: conditions — Skull Base Neoplasms | interventions — Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- endotracheal tube (Active Comparator): Procedure: Endotracheal tube
  Hemodynamic variables (blood pressure, HR, CO, rSO2, TCD) will be recorded at 8 moments:
  * baseline, in the operating room before anesthetic induction (non invasive arterial pressure)
  * end of surgery, before awakening (ETT group) or before ETT replacement (LMA group)
  * at 1, 5, 10, 15, 30 and 60 min after extubation or LMA removal (according to group assignment).
  Interventions: Device: endotracheal tube
- Laryngeal mask (Active Comparator): Procedure: Laryngeal mask
  Hemodynamic variables (blood pressure, HR, CO, rSO2, TCD) will be recorded at 8 moments:
  * baseline, in the operating room before anesthetic induction (non invasive arterial pressure)
  * end of surgery, before awakening (ETT group) or before ETT replacement (LMA group)
  * at 1, 5, 10, 15, 30 and 60 min after extubation or LMA removal (according to group assignment).
  Interventions: Device: Laryngeal mask

INTERVENTIONS:
Device: endotracheal tube — In the Endotracheal group In the ETT group, the procedure will be exactly the same except that the ETT will not be exchanged and the patient will be directly extubated
  Hemodynamic variables (blood pressure, HR, CO, rSO2, TCD) will be recorded at 8 moments:
  * baseline, in the operating room before anesthetic induction (non invasive arterial pressure)
  * end of surgery, before awakening (ETT group) or before ETT replacement (LMA group)
  * at 1, 5, 10, 15, 30 and 60 min after extubation or LMA removal (according to group assignment).
  Arms: endotracheal tube
Device: Laryngeal mask — In the LMA group, after aspirating pharyngeal secretions and with the patient still under general anesthesia, we will insert a Proseal LMA (Laryngeal Mask Co. Ltd., Le Rocher, Victoria, Mahe Seychelles) and extubate the trachea using a guided Bailey technique
  Hemodynamic variables (blood pressure, HR, CO, rSO2, TCD) will be recorded at 8 moments:
  * baseline, in the operating room before anesthetic induction (non invasive arterial pressure)
  * end of surgery, before awakening (ETT group) or before ETT replacement (LMA group)
  * at 1, 5, 10, 15, 30 and 60 min after extubation or LMA removal (according to group assignment).
  Arms: Laryngeal mask

SUMMARY:
The endoscopic endonasal transsphenoidal surgery (EETS) is widely used. Although the incidence of complications is low, hypertensive episodes during surgery and awakening and cerebro spinal fluid (CSF) leakage have been described. The occurrence of coughing or vomiting during the early postoperative period must be avoid to protect the patient from CSF leakage and arterial hypertension. The emergency of anesthesia with laryngeal mask has a better haemodynamic profile and less incidence of cough in some surgical procedures and it could help minimizing the risks after EETS

DETAILED DESCRIPTION:
Randomization

At the end of surgery, the anesthesiologist will open a sealed envelope labeled with software-generated randomized numbers to assign the patients, who will be allocated in a 1:1 ratio from nonstratified blocks of four patients, to one of two groups to emerge from anesthesia with the ETT still in place (ETT group) or after it has been replaced by a LMA (LMA group).

Study procedure

In the LMA group, after aspirating pharyngeal secretions and with the patient still under general anesthesia, the investigators will insert a Proseal LMA (Laryngeal Mask Co. Ltd., Le Rocher, Victoria, Mahe Seychelles) and extubate the trachea using a guided Bailey technique. Specifically, the LMA will be inserted after first advancing a suction catheter along the drain tube 8-10 cm beyond the distal end; the mask will be then inserted using a digital technique behind the orotracheal tube, allowing the suction catheter to enter the esophagus first and guiding the tip of the cuff. A number 4 or 5 mask will be chosen for patients weighing 50-70 kg or 70-100 kg, respectively. The cuff will be inflated to a pressure of 60 cmH2O measured with a manometer. Then the orotracheal tube balloon will be deflated and the tube removed. Ventilation then will be continued with the same parameters as had been used earlier.

Administration of neuromuscular relaxants will be then stopped so the patient could emerge from anesthesia. Once the patient recover 2/4 responses of the TOF, neostigmine (0.03 mg/Kg) and atropine (0.01mg/kg) will be given to reverse the neuromuscular blockade and Target-controlled infusion of anesthetics will be stopped. Lidocaine will not be administrated.

Gentle manual ventilator assistance will be then provided until the patient resume spontaneous breathing and respond to simple commands; the LMA or the ETT, depending on the group, will be then removed.

The investigators will administer prophylaxis of nausea in the postoperative period with ondansetron 4 mg/8h/iv.

In the ETT group, the procedure will be exactly the same except that the ETT will not be exchanged and the patient will be directly extubated when the patient will fulfill the same criteria.

Parameters

Patient variables (age, weight, height, sex) and relevant aspects of past medical history, such as:

* controlled hypertension
* tobacco addiction
* respiratory disease will be also registered, including sleep apnea and any chronic respiratory disease (chronic bronquitis, emphysema, chronic pulmonary obstructive disease).
* cough test

Diagnosis, type of surgery, the placement of lumbar drainage.

Hemodynamic variables (blood pressure, HR, CO, rSO2, TCD) will be recorded at 8 moments:

* baseline, in the operating room before anesthetic induction (non invasive arterial pressure)
* end of surgery, before awakening (ETT group) or before ETT replacement (LMA group)
* at 1, 5, 10, 15, 30 and 60 min after extubation or LMA removal (according to group assignment).

The last blood pressure and HR measurements will be taken in the postoperative recovery room. Respiratory variables (including end-tidal carbon dioxide concentration) will be controlled during MV.

* Neurosurgeon will rate the amount of blood in the surgical field (1: no blood; 2: small bleeding that does not interfere with surgery; 3: bleeding that interferes with surgery but surgery is possible; 4: bleeding that impedes normal development of surgery).
* Any coughing episode during the first 5 minutes of awakening. Considering light coughing (1 cough) and strong coughing (access of cough).
* Preoperative xylometazoline administration.
* Intraoperative hypertension and antihypertensive agent administered.
* Endotracheal tube size and laryngeal mask size.
* Difficulties in LMA ventilation.
* Postoperative nausea or vomiting
* CSF leakage during the admission and in the first month.
* Postoperative bleeding.

The objective of the investigators study is evaluate the incidence of coughing and hypertension during awakening in patients after EETS comparing the effect of laryngeal mask vs orotracheal tube.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo EETS in Hospital Clínic de Barcelona

Exclusion Criteria:

* Re-interventions
* Predicted difficult airway (severe acromegalia, mouth opening reduction) or Cormack-Lehane grade IV detected during laryngoscopy
* Risk of bronchial aspiration (e.g., gastroesophageal reflux disease or lower cranial nerve palsy)
* Uncontrolled arterial hypertension detected during preoperative assessment
* Contraindication for early emergence based on anaesthetic or surgical criteria or as a result of complications developing during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure | changes from baseline systolic blood pressure in the first 60 minutes after extubation
  Changes in systolic blood pressure comparing two methods lma vs ett

SECONDARY OUTCOMES:
noradrenaline levels | changes from baseline noradrenaline level at 30 minutes after awakening
  Compare noradrenaline levels in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Paola Hurtado, MD, Principal Investigator — Senior Especialist
Locations (1):
- Anesthesia department, Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided